CLINICAL TRIAL: NCT03711799
Title: Mind the Gap Intervention
Brief Title: Mind the Gap (AIR-B3)
Acronym: MtG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Collaborators: University of Rochester (Other); University of Pennsylvania (Other); University of California, Davis (Other); Drexel University (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor/PhD, Health Resources and Services Administration (HRSA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-000029
Record Dates: First submitted 2018-10-12; First posted 2018-10-18 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Services; Mind the Gap; Peer Coach
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resource Only Group (No Intervention): Families randomized to the resource only condition will have access to training materials in web-based and paper formats. The will receive the internet address to access web-based trainings, handouts and materials, including instructions for each activity and they will receive a binder that includes the information that is available on line so they can access the information even if they do not have internet access. Families in the resource only condition will not have access to a peer coach through the program. They will not have access to the on-line support community.
- Peer Coaching Group (Experimental): Families randomized to peer coaching will receive assistance with navigating the training program and accessing the system from a trained peer parent coach. Peer coaches will, as much as possible, be culturally and language-matched with the participant family.
  Interventions: Behavioral: Access to services via peer coaching

INTERVENTIONS:
Behavioral: Access to services via peer coaching — This intervention will allow for half of the participants, randomly selected, to get help navigating the system of acquiring services for their child. These participants will be assisted by a coach who are also parents of a child with autism and have already been through the process.
  Arms: Peer Coaching Group

SUMMARY:
There has been a lack of research on the unique needs of families with autism in the African-American and Latino communities. The process of screening, evaluation and treatment for children with autism can be long and arduous, especially in these communities. This often means that the best interventions for children with autism are not reaching minority communities. For many families, the complexity of the services system leads to a long wait after the initial diagnosis before accessing intervention. This means that the children have delayed access to treatment. Mind the Gap is a study that seeks to provide immediate and culturally appropriate support for families who have just received diagnosis but have yet to receive treatment. This support will be provided in families' native languages and, through the use of phone and video sessions, can accommodate busy schedules. Mind the Gap participants will be randomized to receive one of two conditions, which are 1.Resources only (online training modules and paper or on line resource lists, but no peer coaching) 2. Peer coaching (will receive all online training access). The peer coaches will be recruited from local parent support agencies. They will not be professionals in the field of ASD, but they will be trained by the research group on how to access the online tools and how to work whith families. They will contact the participants via phone or video conference on a weekly basis and an in- person visit per month for 3 months. Peer coaches will have a monthly call with participants for an additional nine months.We hope that this study will help the African American and Latino communities receive services sooner than currently reported. We also hope that in the future, parent organizations will use these tools to help families that have recently received an ASD diagnosis will us navigate the complex system of attaining services.

DETAILED DESCRIPTION:
We will recruit 140 (35 per site) families that will be referred by pediatricians, school staff, family resource centers, early intervention agencies, DDS or self-referred using study referral form, phone or web based referral system. The referral will include consent to be contacted by the research team. All families will complete the screening survey by phone (Section 19.2, item 3.1) with a member of the research team. This will be the only survey that will determine eligibility. If eligible to participate, the participants will be asked to give an oral consent. The oral consent will allow the research team to randomize the family to either the Resource Only Group or the Peer Coaching Group. For both conditions, a written consent will be later obtained when the research team meets with the families for the intake survey and filling out the measures: Demographic, Family Empowerment Scale, Caregiver Agency Questionnaire, Caregiver Autism Knowledge Questionnaire, Caregiver Stigma Scale and a Satisfaction Survey only at end of study. Cultural Capital Survey will only be used once at the intake survey meeting.

Parents will have access to ParentSquare, a safe, secure platform for program-to-parent and parent-to-parent communication. ParentSquare has a registration feature where parents can complete forms and sign up for courses and training modules and to broadcast training. Parents can choose to be notified via text, email with reminders or updates through the app. Messages can be private or broadcasted to larger group. There is also a document feature to allow shared access between parent and coach of parent goals and progress between calls and visits. Each site will be responsible for monitoring communication of their participants in Parent Square along with Drexel University.

Participants will also include up to 40 peer coaches (10 per site) who will be trained to provide coaching to families for 5 months as a family gains access to services. Peer Coach Inclusion criteria: (1) parent of a child with autism or other similar developmental disorder; (2) a child over 9 years old and at least 5 years post-diagnosis; (3) some experience working with parents and/or understanding of the service system and (4) fluent in English and/or Spanish.

Intervention Resource only. Families randomized to the resource only condition will have access to training materials in web-based and paper formats. The will receive the internet address to access web-based trainings, handouts and materials, including instructions for each activity and they will receive a binder that includes the information that is available on line so they can access the information even if they do not have internet access Families in the resource only condition will not have access to a peer coach through the program. They will not have access to the on-line support community.

Peer Coaching Condition. Families randomized to peer coaching will receive assistance with navigating the training program and accessing the system from a trained peer parent coach. Peer coaches will, as much as possible, be culturally and language-matched with the participant family. Families in this condition will receive a call from their peer coach who will set up an initial, in-person meeting either in-home, clinic or community setting depending on the participant preference. Based on the goal setting interview the peer coach and the family will choose initial goals to complete in the first week, which will include (1) completion of a training (typically the What is ASD? Training will be completed first); (2) completion of one activity related to service access (e.g., phone access; call to service provider; form completion); and (3) one self-care activity. A timeline for goals will be developed together based on the family needs. Peer coaches will have a guide for rating the importance of training and materials for the family based on the interview, and a guide which will identify triggers (e.g. challenging behavior, safety concerns) to increase the level of care. Peer coaches will set up a weekly call or video conferences (based on parent preference), and monthly in person visit with the family to assess goal progress, provide information, and set up subsequent goals and/or additional support if needed. Monthly visits and weekly calls will continue for 12 visits up to 4 months). If parents choose to meet via video conference, a secure, University approved method will be used by coaches (e.g., Zoom, Skype, Webex). Three of the calls will be audio recorded for research purposes and to provide feedback to the coaches. Calls will then be reduced to monthly for 9 months. Parent participants can contact the peer coach at any time as well. Peer coaches will have a script and materials for each call which will cover a specific topic identified with the family. Peer coaches will have bi monthly supervision.

Peer Coach Training. Peer coaches will be hired or referred from local parent support agencies . Compensation will be specific to each site. Peer coaches are parents of children with ASD diagnosed at least 5 years ago, fluent in English or Spanish and have some experience helping other families of children with ASD.

Peer coaches will attend four, 3-hour training sessions in the use of the intervention materials. They will have a chance to practice using the materials and will learn about issues related to safety and how to work with families. They will complete citi training and additional training and role play in the confidentiality. Training will include learning to use Parentsquare and role playing interviewing and discussing topics with families. Coaches will have access to scripts for each potential topic and resources to address family needs. Parent engagement in the intervention will also be measured by (1) enrollment in sessions; (2) attendance at sessions and peer coach calls/meetings; (3) accessing on-line materials; (4) completion of on-line trainings; and (5) project attrition.

Peer coaches will be expected to provide a 24-hour notice if they need to cancel a meeting or session. They will also be expected to reschedule missed appointments. Also, peer coaches will not be paid for missed appointments. If the peer coaches misses 3 meetings in a row without proper cancellation, a member of the research team will have to resume his/her activities.

ELIGIBILITY:
Parent Inclusion Criteria:

* child under 9 years of age with a diagnosis of ASD
* no receipt of ASD specific services outside of school (family may still qualify if child is connected with a regional center/EI, but not yet receiving services), defined as (a) services obtained through insurance based on having an ASD diagnosis;or (b) receiving services through 0-3 that can only be accessed with an ASD dx (e.g., intensive in home EIBI)
* family income is under 250% of the federal guidelines for poverty rate
* English or Spanish speaking.

Peer Coach Inclusion criteria:

* parent of a child with autism or other similar developmental disorder
* a child over 9 years old and at least 5 years post-diagnosis
* some experience working with parents and/or understanding of the service system and
* fluent in English and/or Spanish.

Parent Exclusion Criteria:

* child is in out-of-home placement or foster care.

Peer Coach Exclusion Criteria:

* Cannot commit to the times and requirements of the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Service Access Form from month to month | Monthly from baseline and up to a year after baseline
  This form was created within the research group. It is used monthly after entry to document the services the participants would like to get and the ones they are currently receiving.

SECONDARY OUTCOMES:
Family Empowerment Scale (Koren, DeChillo & Friesen, 1992) | baseline, 4 months, 8 months and a year after baseline
  It is a 34-item rating scale that measures empowerment in families with children who have emotional, behavioral, or developmental disorders. The FES has three subscales, Family, Service System and, Social Politics. Parents rated each item on a 5-point Likert-type rating scale.
Caregiver Agency Questionnaire (adapted from Kuhn & Carter, 2006) | baseline, 4 months, 8 months and a year after baseline
  It is a 20 item survey about how often the parent engaged in certain activities related to promoting child development. For each question responses are on a Likert scale from 1=never to 5=almost always. Ten questions related to items targeted in the intervention were chosen, with assistance from one of the developers (Dr. Carter).
Caregiver Autism Knowledge Questionnaire (adapted, Kuhn & Carter, 2006) | baseline, 4 months, 8 months and a year after baseline
  It is a 43-item true/false questionnaire that measures knowledge of facts about autism in the areas of diagnosis, symptoms, treatments and interventions, and etiology. To reduce burden we have chosen 10 questions representative of information provided in the intervention and approved by the survey author (Dr. Carter) . Caregivers will respond to each true/false item.
Caregiver Stigma Scale (McKay & Cavaleri, 2009) | baseline, 4 months, 8 months and a year after baseline
  It is an 11-item scale adapted from McKay and Cavaleri (2009) that measures the degree of stigma that caregivers have about receiving professional services or treatment for their child from a mental health or developmental specialist (e.g. developmental pediatrician, psychologist, psychiatrist). Caregivers will utilize a 5-point Likert-type rating scale to rate the extent to which they agreed with statements regarding beliefs about accessing professional services for their child (e.g. "I believe that there is something wrong with children who get professional services or treatment").
Satisfaction Survey | 4 months post baseline
  This survey was created by the research team. At 4 months post entry, caregivers will rate their satisfaction with the intervention on a survey that utilizes a 5-point Likert-type rating scale.
Community Capital Scale | baseline
  This survey measures how each parent's community involvement/importance influences their behavior. It was created by a member of the research group.
Social Dynamics of Intervention_ASD (Autism Spectrum Disorder)-SoDI | baseline, 4 months, 8 months and a year after baseline
  This measure shows the level of support the parent has with his/her child with autism.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC Davis, Davis, California
  - University of Rochester, Rochester, New York
  - UPENN, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Iadarola S, Pellecchia M, Stahmer A, Lee HS, Hauptman L, Hassrick EM, Crabbe S, Vejnoska S, Morgan E, Nuske H, Luelmo P, Friedman C, Kasari C, Gulsrud A, Mandell D, Smith T. Mind the gap: an intervention to support caregivers with a new autism spectrum disorder diagnosis is feasible and acceptable. Pilot Feasibility Stud. 2020 Sep 7;6:124. doi: 10.1186/s40814-020-00662-6. eCollection 2020. PMID 32944273